CLINICAL TRIAL: NCT06294054
Title: Survival prEdiction in bLadder Cancer Patients Treated by nEoadjuvant Chemotherapy Before cysTectomy
Brief Title: Bladder Cancer and Neoadjuvant Chemotherapy Efficiency Before Cystectomy
Acronym: SELECT
Status: Active, not recruiting | Type: Observational
Sponsor: University Hospital, Rouen (Other)
Collaborators: Institut Curie (Other)
Responsible Party: Sponsor
Other Study IDs: 2021/0393/HP
Record Dates: First submitted 2024-02-27; First posted 2024-03-05 (Actual); Last update posted 2024-03-06 (Actual); Status verified 2024-03

CONDITIONS: Bladder Cancer; Genomic Instability
Keywords: Neoadjuvent chemotherapy; Molecular subtype; Bladder cancer; Genomic instability; Artificial intelligence
MeSH Terms: conditions — Urinary Bladder Neoplasms; Genomic Instability | interventions — Neoadjuvant Therapy

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (3):
- Patients enrolled in VESPER study: Tumors from patient having muscle invasive bladder cancer who benefit from neoadjuvant chemotherapy with cisplatine included in VESPER cohort
  Interventions: Combination Product: neoadjuvant chemotherapy with cisplatine
- Patients from St Louis cohort not enrolled in VESPER study: Tumors from patient having muscle invasive bladder cancer who benefit from neoadjuvant chemotherapy with cisplatine included in Saint-Louis cohort
  Interventions: Combination Product: neoadjuvant chemotherapy with cisplatine
- Patients from COBLAnCE cohort not enrolled in VESPER study: Tumors from patient having muscle invasive bladder cancer who benefit from neoadjuvant chemotherapy with cisplatine included in COBLAnCE cohort
  Interventions: Combination Product: neoadjuvant chemotherapy with cisplatine

INTERVENTIONS:
Combination Product: neoadjuvant chemotherapy with cisplatine — Blood from patient having muscle invasive bladder cancer who benefit from neoadjuvant chemotherapy with cisplatine

SUMMARY:
This study will allow the investigators to better assess the efficiency of neoadjuvant chemotherapy before cystectomy by training a predictive model on different patient cohorts with bladder cancer.

DETAILED DESCRIPTION:
The project is based on three prospective cohorts of patients with MIBC: the VESPER trial (n=296), the St-Louis Hospital cohort (n=99), and the COBLAnCE cohort (n=312). Using WES and RNAseq, the investigators will determine genomic instability, DDR gene mutation and molecular subtypes. After digitization of tumour slides, the investigators will train and test predictive models based on deep learning approaches to predict outcome after neoadjuvant chemotherapy, either by estimating molecular subtypes and genetic features from pathological images, or by directly defining a prognostic signature. The statistical analyses will assess the performance of the models combining genomic instability, DNA Damage Response mutations and/or molecular subtyping to predict outcome after neoadjuvant chemotherapy and compare them with the models based on WSI deep learning approaches. These results will help to design new therapeutic strategies.

ELIGIBILITY:
Inclusion Criteria:

- Inclusion Criteria of Patients enrolled in VESPER study:

Blood and tumors from patient having muscle invasive bladder cancer who benefit from neoadjuvant chemotherapy with cisplatine included in VESPER cohort and :

having signed an informed consent form for the participation to the collection or dead/lost to follow-up without prior opposition expressed against research program, genetic analysis will only be carried out for patients who have signed the genetic consent form.

- Inclusion Criteria of Patients from St Louis cohort not enrolled in VESPER study:

Blood and tumors from patient having muscle invasive bladder cancer who benefit from neoadjuvant chemotherapy with cisplatine included in Saint-Louis cohort and :

being informed for the participation to the collection and not having expressed opposition against research program or dead/lost to follow-up without prior opposition expressed against research program,

- Inclusion Criteria of Patients from St Louis cohort not enrolled in COBLaNCE study:

Blood and tumors from patient having muscle invasive bladder cancer who benefit from neoadjuvant chemotherapy with cisplatine included in COBLaNCE cohort and :

being informed for the participation to the collection and not having expressed opposition against research program or dead/lost to follow-up without prior opposition expressed against research program,

Exclusion Criteria:

* Patients not fulfilling eligibility criteria

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: cohorts of patients with MIBC (Muscle-invasive bladder cancer)
Sampling Method: Non-Probability Sample
Enrollment: 707 (Estimated)
Dates: Start 2023-04-01 (Actual); Primary Completion 2026-03-31 (Estimated); Study Completion 2026-03-31 (Estimated)

PRIMARY OUTCOMES:
Progression-free survival | 3 years
  The time from enrollment to progression or death

SECONDARY OUTCOMES:
Overall survival | 5 years
  The time from enrollment to death

CONTACTS AND LOCATIONS:
Overall Officials: Yves ALLORY, MD, Study Director — Institut Curie
Locations (7):
- France (7):
  - Centre de lutte contre le cancer François Baclesse, Caen
  - Centre de recherche des Cordeliers, Paris
  - Hôpital Saint-Louis AP-HP, Paris
  - Institut Curie Centre de Recherche, Paris
  - Institut Curie, Paris
  - Institut Gustave Roussy, Paris
  - Mines ParisTech, Paris

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Background] Pfister C, Gravis G, Flechon A, Soulie M, Guy L, Laguerre B, Mottet N, Joly F, Allory Y, Harter V, Culine S; VESPER Trial Investigators. Randomized Phase III Trial of Dose-dense Methotrexate, Vinblastine, Doxorubicin, and Cisplatin, or Gemcitabine and Cisplatin as Perioperative Chemotherapy for Patients with Muscle-invasive Bladder Cancer. Analysis of the GETUG/AFU V05 VESPER Trial Secondary Endpoints: Chemotherapy Toxicity and Pathological Responses. Eur Urol. 2021 Feb;79(2):214-221. doi: 10.1016/j.eururo.2020.08.024. Epub 2020 Aug 28. PMID 32868138
- [Background] Pfister C, Gravis G, Flechon A, Chevreau C, Mahammedi H, Laguerre B, Guillot A, Joly F, Soulie M, Allory Y, Harter V, Culine S; VESPER Trial Investigators. Dose-Dense Methotrexate, Vinblastine, Doxorubicin, and Cisplatin or Gemcitabine and Cisplatin as Perioperative Chemotherapy for Patients With Nonmetastatic Muscle-Invasive Bladder Cancer: Results of the GETUG-AFU V05 VESPER Trial. J Clin Oncol. 2022 Jun 20;40(18):2013-2022. doi: 10.1200/JCO.21.02051. Epub 2022 Mar 7. PMID 35254888